CLINICAL TRIAL: NCT04473885
Title: Effects of Multi-directional Perturbation-based Balance Training on Postural Control and Cortical Modulation in Elderly With Fall Risk
Brief Title: Effects of Perturbation-based Balance Training on Postural Control and Cortical Modulation in Elderly With Fall Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM109047F
Record Dates: First submitted 2020-07-12; First posted 2020-07-16 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Old Age; Debility; Fall
Keywords: Perturbation-based balance training; Postural control; Cortical modulation; Elderly
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perturbation-based balance training group (Experimental): Participants in the experimental group will receive the balance training under perturbation on Balance SystemTM SD, including limits of stability training, maze control training, random control training. The intervention is 40 min/session, 3 sessions/week for 6 weeks.
  Interventions: Other: Perturbation-based balance training
- Control group (No Intervention): Participants in the control group will remain their regular activity without additional training.

INTERVENTIONS:
Other: Perturbation-based balance training — Participants in the experimental group will receive the balance training under perturbation on Balance SystemTM SD, including limits of stability training, maze control training, random control training. The intervention is 40 min/session, 3 sessions/week for 6 weeks.
  Arms: Perturbation-based balance training group

SUMMARY:
This is a single-blinded randomized controlled trial with pre- and post- measurements. Forty community-dwelling elderly (age> 65 y/o) with fall risk (defined as functional reach test≦25.4 cm) will be recruited and randomly assigned to experimental group or control group (n=20 for each group). Participants in the experimental group will receive the balance training under perturbation on Balance SystemTM SD, including limits of stability training, maze control training, random control training. The intervention is 40 min/session, 3 sessions/week for 6 weeks. Participants in the control group will remain their regular activity without additional training. The primary outcomes include the limit of stability (LOS) of posture control by Balance Master® and brain modulation by Event-Related Desynchronization (ERD) collected by electroencephalogram (EEG). Secondary outcomes include the sensory organization test (SOT), Berg balance scale (BBS), and falls efficacy scale International (FES-I).

DETAILED DESCRIPTION:
Background: Falling is one of the common factors affecting the health in older people. It would cause severe consequences and result in decreasing mobility and independent activity of daily living. According to previous study, balance impairment is the frequent factor for fall in elderly. To maintain balance, reactive postural control ability is the key element from falling. It is suggested that perturbation-based balance training can improve reactive balance performance. However, few studies focus on multi-direction perturbation to mimic the perturbation experienced in daily living. Furthermore, the related cortical activity changes after perturbation-based balance training is not known.

Purpose: The purpose of this study is to explore the effects of multi-directional perturbation-based balance training on posture control and brain modulation in elderly with fall risk.

Methods: This is a single-blinded randomized controlled trial with pre- and post- measurements. Forty community-dwelling elderly (age> 65 y/o) with fall risk (defined as functional reach test≦25.4 cm) will be recruited and randomly assigned to experimental group or control group (n=20 for each group). Participants in the experimental group will receive the balance training under perturbation on Balance SystemTM SD, including limits of stability training, maze control training, random control training. The intervention is 40 min/session, 3 sessions/week for 6 weeks. Participants in the control group will remain their regular activity without additional training. The primary outcomes include the limit of stability (LOS) of posture control by Balance Master® and brain modulation by Event-Related Desynchronization (ERD) collected by electroencephalogram (EEG). Secondary outcomes include the sensory organization test (SOT), Berg balance scale (BBS), and falls efficacy scale International (FES-I). Independent t test and Chi-square test are used for baseline characteristic analysis. All outcomes will be analyzed by repeated measures two-way ANOVA with Tukey post hoc test for within-group and between-group comparisons. Statistical significance is set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 y/o community-dwelling elderly with fall risk (Functional reach test ≦25.4 cm).
* Mini-Mental State Examination score (MMSE) ≧ 24.
* Able to walk independently without assistance at least 10 meters.

Exclusion Criteria:

* With any neurological, mental or cognitive disorders, and orthopedic, pulmonary or cardiac problems that could restrict or preclude their participation in exercise.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Limits of Stability | 15 minutes
  Assessing posture control by Balance Master®
Cortical modulation | 1 hour
  Assessing brain modulation by Event-Related Desynchronization (ERD) collected by electroencephalogram (EEG)

SECONDARY OUTCOMES:
Sensory Organization Test | 15 minutes
  Assessing by Balance Master®
Berg Balance Scale | 15 minutes
  Total score is ranged 0-56, higher scores mean a better outcome.
Falls Efficacy Scale International | 15 minutes
  Total score is ranged 16-64, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, Study Chair — National Yang Ming Chiao Tung University, Taiwan, R.O.C.
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No